CLINICAL TRIAL: NCT02650128
Title: Prospective Multi-Center, Single Arm Study of the Shockwave Coronary Rx Lithoplasty® System in Coronary Arteries
Brief Title: Shockwave Coronary Rx Lithoplasty® Study (Disrupt CAD I)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD 0257
Record Dates: First submitted 2015-12-22; First posted 2016-01-08 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Calcified Coronary Lesions; Coronary Arterial Stenosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lithoplasty System (Experimental): Shockwave Coronary Rx Lithoplasty® System is a lithotripsy-enhanced, low-pressure balloon dilation of calcified, stenotic de novo coronary arteries prior to stent placement
  Interventions: Device: Shockwave Coronary Rx Lithoplasty® System

INTERVENTIONS:
Device: Shockwave Coronary Rx Lithoplasty® System — The Shockwave Coronary Rx Lithoplasty® System is a proprietary balloon catheter system designed to deliver localized, lithotripsy-enhanced, balloon dilatation of calcified, stenotic, de novo coronary arteries. Energizing the lithotripsy electrodes will generate pulsatile mechanical energy within the target treatment site and will disrupt calcium within the lesion and allow subsequent dilatation of a coronary artery stenosis using low balloon pressure. The system consists of a rapid exchange balloon catheter with integrated, internal lithotripsy electrodes and a Shockwave generator.
  Other Names: Coronary Rx Lithoplasty System

SUMMARY:
Prospective, multi-center, single arm study designed to evaluate the safety and performance of the Shockwave Coronary Rx Lithoplasty® System to treat calcified lesions in the coronary arteries for the purpose of enhancing the placement of stents and reducing the ultimate residual stenosis. Patients will be followed through discharge and at 30 and 180 days.

DETAILED DESCRIPTION:
Prospective, multi-center, single arm study designed to evaluate the safety and performance of the Shockwave Coronary Rx Lithoplasty® System to treat calcified lesions in the coronary arteries for the purpose of enhancing the placement of stents and reducing the ultimate residual stenosis. Patients will be enrolled and consented in the study based on history and in some instances an angiogram obtained prior to the study. The study is designed to demonstrate that the Shockwave device can safely and effectively deliver localized shockwave energy for balloon dilatation of calcified, stenotic, coronary arteries. Subjects will be prepared for PCI per the institution's standard protocol. Medications will be administered per the treatment protocol. Femoral access will be obtained using a 6F access sheath, and guiding catheter placed at the ostia of the right or left coronary artery. Baseline angiography of the culprit lesion will be performed prior to placement of a 0.014" guide wire. Baseline and either IVUS or OCT will be performed to determine the Maximum Lumen Area (MLA), percent stenosis, and volumetric lesion assessment. Baseline angiography will be performed to determine lesion length, % stenosis and reference vessel diameter. The investigational device will be prepped per the IFU and positioned at the target lesion. The distal end of the balloon catheter will be connected to the patient cable. The balloon catheter will be inflated to 4 atm and the investigator will deliver 10 pulses for 20 seconds. The balloon will then be inflated to reference vessel diameter and then deflated to reestablish flow and complete one treatment cycle. The treatment cycle will then be repeated. Angiography and either IVUS or OCT will be repeated for the treated lesion.. A coronary stent will be deployed at the site of treatment. Angiography and either IVUS or OCT will be performed following stent placement. Patients will be followed through discharge and at 30 and 180 days. A subset of up to five (5) subjects will receive an angiographic assessment at the 180 day follow up visit, per the Sponsor's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years of age
2. Troponin must be less than or equal to the upper limit of lab normal value within 12 hours prior to the procedure
3. The target vessel must have a TIMI flow 3 at baseline
4. Patients with significant (≥ 50% diameter stenosis) native coronary artery disease including stable or unstable angina and silent ischemia, suitable for PCI
5. Ability to tolerate dual antiplatelet agent (i.e. aspirin, clopidogrel, prasugrel, or ticagrelor for 1 year and single antiplatelet therapy for life
6. Single lesion stenosis of protected LMCA, or LAD, RCA or LCX artery ≥50% in a reference vessel of 2.5 mm - 4.0 mm diameter and ≤ 32 mm length
7. Presence of calcification within the lesion on both sides of the vessel as assessed by angiography
8. Planned treatment of single lesions in one vessel
9. Ability to pass a 0.014" guide wire across the lesion
10. Patient, or authorized representative, signs a written Informed Consent form to participate in the study, prior to any study-mandated procedures
11. Patient is able and willing to comply with all assessments in the study

Exclusion Criteria:

1. Concomitant use of Atherectomy, Specialty balloon, or investigational coronary devices
2. Prior PCI procedure within the last 30 days of the index procedure
3. Patient has planned cardiovascular interventions within 30 days post index procedure
4. Second lesion with ≥50% stenosis in the same target vessel
5. Left ventricular ejection fraction < 40%
6. Patient refusing or not a candidate for emergency coronary artery bypass grafting (CABG) surgery
7. Uncontrolled severe hypertension (systolic BP >180 mm Hg or diastolic BP >110 mm Hg)
8. Severe renal failure with serum creatinine >2.5 mg/dL
9. Untreated pre-procedural hemoglobin <10 g/dL
10. Coagulopathy manifested by platelet count <100,000 or International Normalized ratio (INR) >1.7 (INR is only required in patients who have taken warfarin within 2 weeks of enrollment)
11. Patients in cardiogenic shock
12. Acute myocardial infarction (MI) within the past one (1) month, and/or elevated Troponin-I or T (with concomitant elevation of CPK) at the time of enrollment.
13. History of a stroke or transient ischemic attack (TIA) within 3 months
14. NYHA class III or IV heart failure
15. Active peptic ulcer or upper gastrointestinal (GI) bleeding within 6 months
16. Patients with a life expectancy of less than 1 year
17. Target vessel < 2.4 mm in diameter
18. Target lesion > 32 mm in length
19. Chronic Total Occlusion (CTO)
20. Previous stent procedure within 5 mm of target lesion
21. Angiographic evidence of a target lesion severe dissection prior to Coronary Lithoplasty treatment
22. Unprotected Left Main diameter stenosis ≥ 50%
23. Visible thrombus (by angiography) at target lesion site
24. Target lesion is located in a native vessel distal to anastomosis with a saphenous vein graft or LIMA/RIMA bypass
25. Patient has active systemic infection
26. Patient has connective tissue disease (e.g., Marfan's syndrome)
27. Patient has a hypercoagulable disorder
28. Uncontrolled insulin dependent diabetes
29. Patient has allergy to imaging contrast media for which they cannot be pre-medicated
30. Evidence of aneurysm in target vessel
31. Patient is pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Fajadet, MD, Principal Investigator — Clinic Pastuer
Locations (7):
- Australia (2):
  - Monash Heart, Monash Health, Clayton, Victoria
  - St. Vincent's Hospital, Melbourne, Victoria
- Clinic Pastuer, Toulouse, France
- Thoraxcenter, Erasmus MC, Rotterdam, Netherlands
- Skane University Hospital- Lund, Lund, Sweden
- United Kingdom (2):
  - King's College Hospital, London
  - Royal Brompton Hospital, London

REFERENCES:
- [Derived] Kereiakes DJ, Di Mario C, Riley RF, Fajadet J, Shlofmitz RA, Saito S, Ali ZA, Klein AJ, Price MJ, Hill JM, Stone GW. Intravascular Lithotripsy for Treatment of Calcified Coronary Lesions: Patient-Level Pooled Analysis of the Disrupt CAD Studies. JACC Cardiovasc Interv. 2021 Jun 28;14(12):1337-1348. doi: 10.1016/j.jcin.2021.04.015. Epub 2021 May 3. PMID 33939604
- [Derived] Brinton TJ, Ali ZA, Hill JM, Meredith IT, Maehara A, Illindala U, Lansky A, Gotberg M, Van Mieghem NM, Whitbourn R, Fajadet J, Di Mario C. Feasibility of Shockwave Coronary Intravascular Lithotripsy for the Treatment of Calcified Coronary Stenoses. Circulation. 2019 Feb 5;139(6):834-836. doi: 10.1161/CIRCULATIONAHA.118.036531. No abstract available. PMID 30715944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment and enrollment took place at seven clinical sites in Australia and Europe between December 2015 and September 2016. A total of 60 subjects with calcified, stenotic de novo coronary arteries were enrolled and treated with the investigational device.
Groups:
- Shockwave Coronary Rx Lithoplasty System: Shockwave Coronary Rx Lithoplasty® System is a lithotripsy-enhanced, low-pressure balloon dilation of calcified, stenotic de novo coronary arteries prior to stent placement
  Shockwave Coronary Rx Lithoplasty® System: The Shockwave Coronary Rx Lithoplasty® System is a proprietary balloon catheter system designed to deliver localized, lithotripsy-enhanced, balloon dilatation of calcified, stenotic, de novo coronary arteries. Energizing the lithotripsy electrodes will generate pulsatile mechanical energy within the target treatment site and will disrupt calcium within the lesion and allow subsequent dilatation of a coronary artery stenosis using low balloon pressure. The system consists of a rapid exchange balloon catheter with integrated, internal lithotripsy electrodes and a Shockwave generator.
Period: Overall Study
Arm/Group | Shockwave Coronary Rx Lithoplasty System
Started | 60
30 Day Primary and Safety Endpoint | 60
Completed (180 day major adverse cardiac event (Post-Market Clinical Follow-up)) | 58
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Shockwave Coronary Rx Lithoplasty System
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 47
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 4
  Sweden | 1
  United Kingdom | 29
  Australia | 16
  France | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety - Frequency of Major Adverse Cardiac Events (MACE) Within 30 Days of the Procedure.
Description: MACE defined as:
  * Cardiac death
  * Myocardial Infarction - defined as a CK-MB level > 3 times the upper limit of lab normal (ULN) value with or without new pathologic Q wave
  * TVR - defined as revascularization at the target vessel (inclusive the target lesion) after the completion of the index procedure
Time Frame: 30 days
Population: No imputation of or adjustments for missing data were performed for the primary analyses. The population for all analysis was the Intent-To-Treat (ITT) analysis set. ITT was defined as those subjects who had insertion of the Lithoplasty catheter attempted, defined as the point of enrollment.
Measure: Number; unit: events
Arm/Group | Shockwave Coronary Rx Lithoplasty System
Number analyzed (Participants) | 60
events | 57

2. Primary Outcome: Performance
Description: The ability of the Shockwave System to produce acceptable residual stenosis (<50%) after stenting with no evidence of in-hospital MACE.
  Clinical success measured by each patient that achieves both these requirements.
Time Frame: Post-procedure (within 24 hours following procedure and prior to discharge)
Population: No imputation of or adjustments for missing data were performed for the primary analyses. The population for all analysis was the Intent-To-Treat (ITT) analysis set. ITT was defined as the subjects who had insertion of the Lithoplasty catheter attempted, defined as the point of enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Coronary Rx Lithoplasty System
Number analyzed (Participants) | 60
Participants | 57

3. Secondary Outcome: Quantitative Assessment of the Residual Stenosis in Treated Lesions
Description: Angiographic success defined as success in facilitating stent deliver with <50% residual stenosis and without serious angiographic complications. Serious angiographic complications defined as severe dissection (Type D to F), perforation, abrupt closure, and persistent slow flow or persistent no reflow
Time Frame: Post-procedure (within 24 hours following procedure and prior to discharge)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Coronary Rx Lithoplasty System
Number analyzed (Participants) | 60
Participants | 58

4. Secondary Outcome: 180 Day MACE
Description: as for outcome 1
Time Frame: 180 days post-procedure
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Lithoplasty System
Number analyzed (Participants) | 58
events | 58

ADVERSE EVENTS:
Time Frame: through 30 days and 6 months
Arm/Group | Shockwave Coronary Rx Lithoplasty System
All-Cause Mortality (participants affected / at risk) | 2/60
Serious Adverse Events (participants affected / at risk) | 10/60
Other Adverse Events (participants affected / at risk) | 37/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shockwave Coronary Rx Lithoplasty System (N=60)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina Unstable (Cardiac disorders) | 1 (1)
Coronary Artery Dissection (Cardiac disorders) | 3 (3)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Cerebral Hypoperfusion (Nervous system disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shockwave Coronary Rx Lithoplasty System (N=60)
Bradycardia (Cardiac disorders) | 1 (1)
Coronary Artery Dissection (Cardiac disorders) | 12 (12)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oesophageal Pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest Discomfort (General disorders) | 2 (2)
Chest Pain (General disorders) | 5 (5)
Puncture Site Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 2 (2)
Enzyme Level Increased (Investigations) | 7 (7)
Troponin Increased (Investigations) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Sciatica (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No